CLINICAL TRIAL: NCT03606291
Title: A Phase II Open-Label Multi-center Trial of Isotoxic Hypofractionated Radiotherapy for NSCLC
Brief Title: NSCLC Isotoxic Hypofractionated Radiotherapy
Acronym: IHR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Xue Xiaoying, Director of Radiotherapy, The Second Hospital of Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC isotoxic HypoRT
Record Dates: First submitted 2018-06-27; First posted 2018-07-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: isotoxic; hypofractionation; Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- isotoxic hypofractionation group (Experimental): 1. Hypofractionated radiation: 3Gy/f. 2,Individualized prescriptions for different patients:
  (1) Spinal cord: 0%>45 Gy, and ≤2 Gy each time Lung: V20≤30%, V5≤65%, MLD≤16Gy Esophagus: highest dose ≤ 72Gy 3. Maximum limit: If the limit of any "A" is not reached, the maximum radiation dose is 72 Gy. The lowest radiation dose: 45Gy.
  Interventions: Radiation: isotoxic hypofractionation

INTERVENTIONS:
Radiation: isotoxic hypofractionation — the normal tissue limits are uniform, such as: V20% ≤ 30%, spinal cord 0> 45Gy, etc., and used hypofractionated radiotherapy technology so that each patient received the maximum individualized radiation dose as possible

SUMMARY:
Radiotherapy plays an important role in non-small cell lung cancer (NSCLC), and concurrent chemoradiation is considered to be the standard treatment for locally advanced NSCLC. However, due to the patient's physical condition, comorbidities and other reasons, only about 1/3 of patients can receive concurrent chemoradiation. Radiotherapy alone or sequential chemoradiation has become the treatment protocol for most patients. Hypofractionated radiotherapy can be used in NSCLC because it can shorten the over treatment time and may potentially reduce the effect of accelerated repopulation and obtain higher biological effective dose（BED）.So far, the vast majority of radiotherapy prescriptions have given a uniform dose of 60 Gy. This unified prescription dosage approach is completely inconsistent with the concept of precision treatment. The Netherlands MAASTRO put forward the concept of in silico radiotherapy prescription, that is: the normal tissue limits are uniform, such as: V20% ≤ 30%, spinal cord 0> 45Gy, etc., This radiation prescription could reach the limits of the normal tissue of every patient; if no one tissue limits were reached, the highest dose was set up to 79.2 Gy (1.8 Gy, BID). MAASTRO applied this "iso-toxic" radiotherapy prescription and used accelerated hyperfractionation technology so that each patient received the maximum individualized radiation dose as possible. We will integrate this concept with hypofractionated radiotherapy in order to further improve patient survival.

DETAILED DESCRIPTION:
Radiotherapy plays an important role in non-small cell lung cancer (NSCLC), and concurrent chemoradiation is considered to be the standard treatment for locally advanced NSCLC. However, due to the patient's physical condition, comorbidities and other reasons, only about 1/3 of patients can receive concurrent chemoradiation. Radiotherapy alone or sequential chemoradiation has become the treatment protocol for most patients. Hypofractionated radiotherapy can be used in NSCLC because it can shorten the over treatment time and may potentially reduce the effect of accelerated repopulation and obtain higher biological effective dose（BED） So far, the vast majority of radiotherapy prescriptions have given a uniform dose of radiotherapy to all patients, regardless of individual factors such as tumor size, location, and adjacent vital organs, which may cause two consequences: First, small-volume tumors may, not receive enough radiation dose, resulting in a decrease in local control rates. Second, for large volumes of tumors or tumors adjacent to vital organs, even the "so-called standard dose" (60 Gy) may cause serious damage to normal tissues. This unified prescription dosage approach is completely inconsistent with the concept of precision treatment. The Netherlands MAASTRO put forward the concept of in silico radiotherapy prescription, that is: the normal tissue limits are uniform, such as: V20% ≤ 30%, spinal cord 0> 45Gy, etc., and each patient receives a different dose of radiation therapy. This radiation prescription could reach the limits of the normal tissue of every patient; if no one tissue limits were reached, the highest dose was set up to 79.2 Gy (1.8 Gy, BID). MAASTRO applied this "iso-toxic" radiotherapy prescription and used accelerated hyperfractionation technology so that each patient received the maximum individualized radiation dose as .From the model study to the long-term survival results, a series of encouraging results were achieved. The use of an individualized radiotherapy prescription based on iso-toxicity for the treatment of NSCLC in large-segment radiotherapy is expected to achieve: 1. For patients with small tumor volumes and no adjacent to vital organs, a higher radiation dose is given under safe conditions. 2. For patients with larger volumes of tumors or adjacent to vital organs, give safer doses.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological or cytological diagnosis of non-small cell lung cancer patients, the clinical stage using the eighth edition of American Joint Committee on Cancer（AJCC）, including stage III without resectable or who when SBRT/SABR are not suitable;
2. Age ≥ 18 years;
3. The expected survival period is ≥ 3 months;
4. KPS score ≥ 60;
5. Normal blood count,liver and kidney function ≤ 2.5 times the upper limit of normal;

Exclusion Criteria:

1. Serious medical problems require hospitalization, included (but not limited to ): history of pulmonary fibrosis, previous myocardial infarction within 6 months, heart failure grade II and above, uncontrolled heart failure, uncontrolled COPD, uncontrolled diabetes Wait;
2. Esophageal invasion (cT4);
3. Others are not suitable for receiving radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
radiation induced esophagitis and radiation induced pneumonitis | 2 years
  Number of participants with treatment-related severe adverse events：Grade IV radiation esophagitis, Grade III radiation esophagitis which results in interruption of radiotherapy for 7 days or more and Grade III or above radiation pneumonitis

SECONDARY OUTCOMES:
TTP | 5 years
  Record the time from the start of enrollment to the objective progression of the tumor
PFS | 5 years
  Record the time from the start of enrollment to the progression of disease or death
OS | 5 years
  Record the time from the start of enrollment to death(for any reason)
LC | 5 years
  Record the time from the start of enrollment to progression or primary tumors

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ying Xue, Professor, Study Director — The Second Hospital of Hebei Medical University; Qiang Lin, Professor, Study Director — North China Petroleum Bureau General Hospital, Hebei Medical University; Chao-Xing Liu, Professor, Study Director — No.1 Hospital of Shijiazhuang City
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No